CLINICAL TRIAL: NCT03519152
Title: To Compare Efficacy of Low Dose Diclofenac (25mg) in Management of Postoperative Pain After Periodontal Flap Surgery: A Clinical Trail.
Brief Title: To Compare Efficacy of Low Dose Diclofenac (25mg) in Management of Postoperative Pain After Periodontal Flap Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr.Kshitij .K. Karmkar, Principle investigator, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: tatyasaheb kore dental college
Record Dates: First submitted 2017-02-01; First posted 2018-05-08 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Diclofenac; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant
Masking Description: patient were masked for which tablet they were reciving during the study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group one side (Experimental): All patients were scheduled for open flap debridement surgery on at least two quadrants ≥1 weeks apart.One group will receive Low Dose Diclofenac tablets (25mg Diclofeanc and 325 mg paracetamol), BID for 3 days. The patients who are diagnosed with generalized moderate/severe chronic periodontitis will be included in study. For each quadrant, a flap was raised under local anesthesia (2% lignocaine with 1:80,000 epinephrine). In both the quadrants same technique of anesthesia will be employed. The location and the extent of surgery, volume of the local anesthesia given, and time required to perform the surgical procedure will be recorded in the patient file. Patients will be instructed to complete a pain diary chart for 3 days.
  Interventions: Drug: low dose diclofenac
- study group second side (Placebo Comparator): Other group will receive Diclofeanc (50mg Diclofenac and 325mg paracetamol), BID for 3 days. The patients who are diagnosed with generalized moderate/severe chronic periodontitis were included in study. For each quadrant, aperiodontal flap was raised under local anesthesia (2% lignocaine with 1:80,000 epinephrine). In both the quadrants same technique of anesthesia will be employed. The location and the extent of surgery, volume of the local anesthesia given, and time required to perform the surgical procedure was recorded in the patient file. Patients were instructed to complete a pain diary chart for 3 days.
  Interventions: Drug: low dose diclofenac

INTERVENTIONS:
Drug: low dose diclofenac — it is a split mouth design in which one side recieved low dose diclofenac(25mg) after periodontal flap surgery and in next week second side will recieve diclofenac 50mg after flap surgery.
  Other Names: periodontal flap surgery; scaling and root planning

SUMMARY:
Pain after periodontal surgical procedures is a common manifestation. The perception of pain is highly subjective and varies substantially among individuals. Many factors affect pain perception, such as the nature, duration, and extent of the surgery and psychological aspects (e.g., stress and anxiety). Pain after periodontal surgery is an example of acute dental pain of mild to moderate severity. Non-steroidal anti-inflammatory drugs (NSAIDs) have a significant advantage in the control of pain after periodontal or oral surgical procedures.

Diclofenac is a powerful anti-inflammatory and analgesic drug that is well suited for local use in the oral cavity. Diclofenac competes with arachidonic acid in a dose dependent manner for binding with platelet COX. This results in decreased production of PG and thus reduces inflammation, swelling and pain.

As Diclofenac associated with many adverse effects, like gastric irritability, nausea, headache, dizziness. Undesirable effects may be minimized by using the lowest effective dose for the shortest duration necessary to control symptoms. As many of clinical trials have suggested Diclofeanc 50 mg alleviates the postoperative pain. So main aim of the study was to evaluate the effectiveness of low dose Diclofenac(25mg) in reducing the post operative pain after periodontal flap surgeries. Thus comparing the effects of low dose Diclofenac and Diclofenac 50mg for reducing post-operative pain.

DETAILED DESCRIPTION:
The present split mouth, single blind randomized controlled clinical trial was carried out in the

Department of Periodontology and source of the patients was from the outpatient section of Tatyasaheb Kore Dental College & Research Centre, New Pargaon.

Patients were enrolled in the study between November 2016 and June 2017. Based ' on the power of study that was l 80% with alpha of 0.05 with SD of ±1.47, we required

18 experimental quadrants and 18 control quadrants. Considering 10% dropout " sample size was finalized at 20.

The study included 20 patients [14 males and 6 females] with generalized chronic periodontitis.

With age ranging from 17-55 years, the selected patient had atleast 20 natural teeth, and with no history of previous periodontal therapy preceding six months of study. Medically compromised patients, pregnant and lactating mothers, smokers and alcoholics, and those with a history of taking anticoagulant therapy, patient reporting intake of steroidal or non-steroidal antiinflammatory drugs (previous 3 months) or antibiotics in previous six month were excluded from the study. Patient with known hypersensitivity to Diclofenac and gastric diseases were also not considered.

The protocol of the study was explained to each patient, and informed consent was obtained after explanation of the study. A split mouth design was used. A total of 40 quadrants in 20 patients (two quadrants in each patient) were operated. Complete medical evaluations of all the patients were done to rule out any systemic conditions.

All patients were scheduled for open flap debridement surgery on at least two quadrants >1 weeks apart. Each quadrant was randomly allocated (coin test) a different medication regimen for postoperative pain control. So in one patient two quadrant were operated one quadrant received Low Dose Diclofenac tablets (25mg Diclofenac and 325 mg paracetamol), BID for 3 days, whereas the other operated quadrant received Diclofenac (50mg Diclofenac and 325mg paracetamol), BID for 3 days.

A flap was raised under local anesthesia (2% lignocaine with 1:80,000 epinephrine). In both the quadrants same technique of anesthesia was employed. The location and the extent of surgery, volume of the local anesthesia given, and time required to perform the surgical procedure was noted in the patient file (Table/Fig 4). Participants were instructed to complete VAS chart once in the morning and once in evening for 3 days with the gap of 8 hours in between and recalled on 4thday and asked about any discomfort noted during following postoperative dayss in the form of questionnaire [Table/fig 5]. For measuring the clinical pain intensity the participants were provided with the visual analog scale (VAS). The VAS consists of a 10-cm line anchored by two extremes: no pain and pain that could not be more severe.

Participants were asked to make a mark on the line representing their level of perceived pain.

STATISTICAL ANALYSIS:- Data were analyzed using statistical software. The P value was set at 0.05 for all tests. The postsurgical pain parameters were presented as mean - SD and were compared using the independent t test.

While for the intra group analysis repeated measures of analysis of variance (ANOVA) test was used and data were presented as mean.

ELIGIBILITY:
Inclusion Criteria:

1. Generalized moderate/severe chronic periodontitis
2. The probing depth (PD) of the surgical sites in the both group ranged from 5 to 8 mm.
3. The clinical attachment level (CAL) at the surgical sites in both the group ranged from 5 to 9 mm.
4. Quadrant with the presence of atleast 6 teeth will be selected for study.

Exclusion Criteria:

1. Tobacco in any form and alcoholics.
2. Pregnant and lactating mother.
3. Patients with history of systemic ailments, patients under ant-inflammatory/antibiotic 3 months prior to recruitment for study.
4. Subjects who had received periodontal treatment within the previous 6 months.
5. Patient who have history of intolerance or hypersensitivity to Diclofenac and with gastric diseases

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-20 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-05-21 (Actual)

PRIMARY OUTCOMES:
visual analog scale VAS | 3 days
  it messures pain intensity it is an 10cm line anchored by two extremes 0 for no pain and 10 for extreme pain

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Khambete, MDS, Study Chair — tatayasaheb kore dental college and hospital new pargaon
Locations (1):
- Dental, Kolhāpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No